CLINICAL TRIAL: NCT06426342
Title: Development and Feasibility of a Metaverse-based Blended Online Intervention to Prevent Employees' Depression: Applying Intervention Mapping
Brief Title: Development and Feasibility of a Metaverse-based Blended Online Intervention to Prevent Employees' Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Suk-Sun Kim, PhD. MSN. RN, Professor, Ewha Womans University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Mindguide_Employee
Record Dates: First submitted 2024-05-14; First posted 2024-05-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-02

CONDITIONS: Depression and Suicide Ideation
Keywords: depression; Employee; Preventive Health Program; Digital Health; Suicide
MeSH Terms: conditions — Depression; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindguide_employee (Experimental)
  Interventions: Behavioral: metaverse-based blended online intervention

INTERVENTIONS:
Behavioral: metaverse-based blended online intervention — A new metaverse-based blended online intervention was developed using an online program and coaching via metaverse to prevent depression among Generation MZ Employees in South Korea.

SUMMARY:
The goal of this feasibility study is to develop a new metaverse-based blended online intervention using an online program and coaching via metaverse to prevent depression among Generation MZ Employees in South Korea. In addition, this study primarily explores reach and acceptability and secondarily evaluates the preliminary effectiveness of this preventive intervention on Korea's Gen MZ Employees.

ELIGIBILITY:
Inclusion Criteria:

* Generation MZ Employees of South Korea who are aged between 20 and 42; Millennials were born between 1981 to 1996, and Generation Zs were born between 1997 to 2004

Exclusion Criteria:

* 1) being unemployed or having less than 1 year job experience,
* 2) having mental disorders such as schizophrenia or substance abuse (as this is a preventive intervention) and currently attending other mental health therapy to avoid mixing effects.

Ages: 20 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Recruitment | baseline
  Recruitment will be assessed by the number of potentially eligible participants enrolled.
The retention rate | Baseline, at 5 weeks after intervention.
  The retention rate will be calculated as the percentage of completion rates for the entire intervention and questionnaires until the completion of a 5 weeks after intervention.
Acceptability | at 5 weeks after intervention.
  Acceptability refers to how participants perceive and feel about the intervention and its components. A 13- item questionnaire was developed based on the Client Satisfaction Questionnaire to measure acceptability with three subcategories: helpfulness (three items), suitability (seven items), and satisfaction (three items). Participants responded on a 5- point Likert scale ranging from 1 (not at all) to 5 (very).

SECONDARY OUTCOMES:
Depression scale | Baseline, at 5 weeks after intervention.
  The Center for Epidemiological Studies Depression Scale with 20- item will be used to measure depressive symptoms using a 4- point Likert scale. The total score ranges from 0 to 60, with higher scores indicating higher levels of depressive symptoms.
Positive and Negative Affect Schedule | Baseline, at 5 weeks after intervention.
  Positive and Negative Affect Schedule will used to measure positive and negative affect using a 5- point Likert scale. The total score ranges from 10 to 50, with higher scores indicating a greater perception of positive affect or negative affect.
Satisfaction with Life Scale | Baseline, at 5 weeks after intervention.
  the Satisfaction with Life Scale with 5- items will be used to assess life satisfaction using a 7- point Likert scale. The total score ranges from 5 to 35, with higher scores indicating greater life satisfaction.
Sleep Quality scale | Baseline, at 5 weeks after intervention.
  Pittsburgh Sleep Quality Index with 19 items will be used to evaluate overall sleep quality. 19 self-reported items includes seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep effi ciency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
  The total score ranges from 0 to 21, with higher scores indicating worse sleep quality.
Burnout assessment tool | Baseline, at 5 weeks after intervention.
  Burnout assessment tool with 23 items will be used to measure burnout including four core burnout symptoms: Exhaustion, Mental Distance, Emotional Impairment, and Cognitive Impairment.
  For each core scale, the average score is calculated by summing the scores of the items in that scale and dividing by the number of items in that scale.
  Score Interpretation:
  1.0 to 1.9: Very low or no burnout symptoms. 2.0 to 2.9: Mild burnout symptoms. 3.0 to 3.9: Moderate burnout symptoms. 4.0 to 5.0: Severe burnout symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Sun Kim, PhD, Principal Investigator — Ewha Womans Univeristy
Locations (1):
- Ewha Womans University, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No